CLINICAL TRIAL: NCT05589103
Title: Mild Head Trauma in the Emergency Room: Assessment of the Risk of Intracranial Hemorrhage in Patients Receving Platelet Inhibitors.
Acronym: Trauma-Head
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7409
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Head Trauma Injury
Keywords: Head Trauma Injury; Head Trauma; Traumatic Intracranial Hemorrhage; Antiaggregants, Platelet
MeSH Terms: conditions — Craniocerebral Trauma; Intracranial Hemorrhage, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical signs presented by a patient with a mild head injury are highly variable but remain strongly predictive of brain damage. The reference examination for the diagnosis of post-traumatic intracranial hemorrhage is currently the cerebral scanner without injection of contrast medium. Magnetic resonance imaging (MRI) tends to surpass CT in equipped centers, except for suspected bone lesions. The time required to perform brain imaging depends on the patient's clinical condition, comorbidities and treatments.

The responsibility of antiplatelet agents in post-traumatic intracranial hemorrhage is currently discussed, particularly with aspirin.

The hypothesis is that there is no significant difference in the proportion of intracranial hemorrhage in patients on antiplatelet agents after mild head trauma, in the absence of other factors favoring the occurrence of intracranial hemorrhage.

ELIGIBILITY:
Inclusion criteria

* Adult patient (≥18 years old)
* Visit to the emergency room of the Strasbourg University Hospital during 2017
* Victim of mild head trauma
* Patient who has given their consent to the reuse of their data for the purposes of this research.

Non-inclusion criteria

* Patient who expressed their opposition to participating in the study
* Subject under safeguard of justice
* Subject under guardianship or curatorship
* Patient on anticoagulant
* Non-isolated head trauma (AVP, fall greater than 6 meters, etc.)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) victim of mild head trauma visiting the emergency room of the Strasbourg University Hospital during 2017.
Sampling Method: Non-Probability Sample
Enrollment: 1692 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Propensity score on the factors influencing the taking of antiplatelet agents. | Files analysed retrospectively from January 01, 2017 to December 31, 2017 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'accueil des urgences - CHU de Strasbourg - France, Strasbourg, France